CLINICAL TRIAL: NCT04041895
Title: Detecting Mild Cognitive Impairment and Probable Alzheimer's Disease From Speech Using Linguistic Deficits With Amyloid PET Imaging as a Baseline.
Brief Title: Detecting Probable Alzheimer's Disease From Speech Using Linguistical Analysis
Status: Withdrawn | Type: Observational
Why Stopped: Unsuccessful in recruiting participants for that study because we needed subjects who had performed Amyloid PET imaging in the last year
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, Sylvester Olubolu Orimaye, Research Associate in the College of Public Health, East Tennessee State University
Other Study IDs: 0218.16sw
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's Disease; Dementia; Linguistics
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's Disease: Those individuals who possess a significant amyloid burden per results of a previous amyloid PET scan radiology report.
  Interventions: Other: Audio speech recording
- Control: Those individuals who do not possess a significant amyloid burden per results of a previous amyloid PET scan radiology report.
  Interventions: Other: Audio speech recording

INTERVENTIONS:
Other: Audio speech recording — Audio recording of speech sample from subject description of Cookie-Theft image.

SUMMARY:
The object of this study is to investigate the use of linguistic deficits from speech samples for the early detection of Mild Cognitive Impairment and probable Alzheimer's disease. It will also evaluate whether the result of the Amyloid PET scan would confirm the effectiveness of a less expensive and less intrusive diagnostic technique through speech

DETAILED DESCRIPTION:
This study will investigate the use of linguistic deficits through a computational diagnostic model for the prediction of Mild Cognitive Impairment (MCI) and Probable Alzheimer's disease (PrAD) from speech samples (verbal utterances). The premise is that MCI and PrAD are characterized by the deterioration of nerve cells that control cognitive speech and language processes, which consequently affects how patients compose verbal utterances. As the Amyloid Positron Emission Tomography (PET) scan is making advances in giving confirmatory evidence of the existence of plaques in the brain, there is the opportunity to investigate whether the result of the scan would confirm the effectiveness of a less expensive and less intrusive diagnostic technique. In this study, participants of a previous IRB approved study on Imaging Dementia-Evidence for Amyloid Scanning (IDEAS) who consent to participate in the new study will be requested to perform a basic descriptive task. The main task to be done by the participants is to verbally describe the scenes on a projected image, while their verbal utterances will be recorded via an audio recorder. The descriptive task is expected to take between 10 to 15 minutes on average. Participants will be required to describe the scenes on the projected Cookie-Theft image (http://www.amyspeechlanguagetherapy.com/thecookie- theft-picture.html). The image is part of the Provide a brief but thorough description of the study. What is the study about? This does not need to contain a summary of background literature. It should just summarize the study itself. Boston Diagnostic Aphasia Examination (BDAE-3) and it is adapted in our study for the purpose of capturing the complexity in the linguistic expression similar to the DementiaBank project (https://talkbank.org/media/DementiaBank/Pitt/cookie/). Note that we are NOT conducting any psychological examination using the BDAE-3, we have only referenced the source of the Cookie-Theft image, which is publicly available for research and has been used for decades. An example of the task is demonstrated in this video: https://www.youtube.com/watch?v=1NB8wBBguMg. The transcripts of the recorded interview will be analyzed by our proposed computational model to detect the presence of Mild Cognitive Impairment or probable Alzheimer's disease. Finally, the IDEAS study PET scan data would be used in conjunction with the transcripts of the recorded interview to compare the results of the linguistic analysis of the transcript with those of the PET scan in making Mild Cognitive Impairment or probable Alzheimer's Disease diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have undergone the Mini Mental State Examination (MMSE).
* Participants who have undergone Amyloid PET scan with a diagnosis of having the Amyloid plaques or not.
* Participants with moderate or fluent English speaking ability.

Exclusion Criteria:

* Participants who cannot speak as the data collection process needs to obtain speech samples.
* Participants who are severely demented or at a very late stage of Alzheimer's disease.
* Participants with stroke.
* Participants who report a history of other neurodegenerative disorders than MCI and AD.
* Participants with chronic vision impairment or who cannot see with the aid of corrective glasses.
* Participants who cannot speak English.
* A participant who have been diagnosed with HIV/AIDS as this may have a cognitive effect on its own.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants would have undertaken an Amyloid PET scan to confirm the presence or absence of Amyloid plaques in the brain through a previously approved study on Alzheimer's disease with Amyloid PET imaging or at the request of their physician to determine possible cause of suspected cognitive decline.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Analysis of speech audio recording describing the "Cookie-Thief Image" using proposed computational model designed by PI for determination of Alzheimer's disease | through study completion, an average of 1 year
  Analysis of speech audio recording of participants description of Cookie-Thief Image The image is part of the Provide a brief but thorough description of the study. What is the study about? This does not need to contain a summary of background literature. It should just summarize the study itself. Boston Diagnostic Aphasia Examination (BDAE-3) and it is adapted in our study for the purpose of capturing the complexity in the linguistic expression similar to the DementiaBank project (https://talkbank.org/media/DementiaBank/Pitt/cookie/) using proposed computational model for determination of Alzheimer's disease

SECONDARY OUTCOMES:
MMSE | through study completion, an average of 1 year
  Mini Mental State Examination

CONTACTS AND LOCATIONS:
Overall Officials: Sylvester O Orimaye, PhD, MPH, Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orimaye, S. O., Wong, J. S. M., & Golden, K. J. (2014, June). Learning predictive linguistic features for Alzheimer's disease and related dementias using verbal utterances. In Proceedings of the 1st Workshop on Computational Linguistics and Clinical Psychology (CLPsych) (pp. 78-87). sn.
- [Background] Orimaye SO, Wong JS, Golden KJ, Wong CP, Soyiri IN. Predicting probable Alzheimer's disease using linguistic deficits and biomarkers. BMC Bioinformatics. 2017 Jan 14;18(1):34. doi: 10.1186/s12859-016-1456-0. PMID 28088191
- [Background] Roark B, Mitchell M, Hosom JP, Hollingshead K, Kaye J. Spoken Language Derived Measures for Detecting Mild Cognitive Impairment. IEEE Trans Audio Speech Lang Process. 2011 Sep 1;19(7):2081-2090. doi: 10.1109/TASL.2011.2112351. PMID 22199464
- [Background] Fraser KC, Meltzer JA, Graham NL, Leonard C, Hirst G, Black SE, Rochon E. Automated classification of primary progressive aphasia subtypes from narrative speech transcripts. Cortex. 2014 Jun;55:43-60. doi: 10.1016/j.cortex.2012.12.006. Epub 2012 Dec 21. PMID 23332818
- [Background] Prud'hommeaux E, Roark B. Graph-Based Word Alignment for Clinical Language Evaluation. Comput Linguist Assoc Comput Linguist. 2015 Dec;41(4):549-578. doi: 10.1162/coli_a_00232. Epub 2015 Dec 1. PMID 34334943
- [Background] Verma M, Howard RJ. Semantic memory and language dysfunction in early Alzheimer's disease: a review. Int J Geriatr Psychiatry. 2012 Dec;27(12):1209-17. doi: 10.1002/gps.3766. Epub 2012 Feb 1. PMID 22298328
- [Background] Reilly J, Rodriguez AD, Lamy M, Neils-Strunjas J. Cognition, language, and clinical pathological features of non-Alzheimer's dementias: an overview. J Commun Disord. 2010 Sep-Oct;43(5):438-52. doi: 10.1016/j.jcomdis.2010.04.011. Epub 2010 May 6. PMID 20493496
- [Background] Klimova B, Maresova P, Valis M, Hort J, Kuca K. Alzheimer's disease and language impairments: social intervention and medical treatment. Clin Interv Aging. 2015 Aug 27;10:1401-7. doi: 10.2147/CIA.S89714. eCollection 2015. PMID 26346123
- [Background] Fraser KC, Meltzer JA, Rudzicz F. Linguistic Features Identify Alzheimer's Disease in Narrative Speech. J Alzheimers Dis. 2016;49(2):407-22. doi: 10.3233/JAD-150520. PMID 26484921
- [Background] 10. Lunsford, R., & Heeman, P. A. (2015, September). Using linguistic indicators of difficulty to identify mild cognitive impairment. In INTERSPEECH (pp. 658-662).

DOCUMENTS (1):
  • Informed Consent Form (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT04041895/ICF_000.pdf